CLINICAL TRIAL: NCT04090151
Title: The RESPOND Outcomes Study - A Study in the RESPOND Consortium (RESPOND: International Cohort Consortium of Infectious Diseases)
Brief Title: The RESPOND Outcomes Study
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Gilead Sciences (Industry); ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Jens D Lundgren, MD, MD, DMSc Professor, Rigshospitalet & University of Copenhagen, Director, CHIP - Centre of Excellence for Health, Immunity and Infections, Rigshospitalet, Denmark
Other Study IDs: The RESPOND Outcomes Study
Record Dates: First submitted 2019-08-30; First posted 2019-09-16 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: HIV
Keywords: HIV; Prospective; Cohort; HCV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (17):
- Austrian HIV Cohort Study (AHIVCOS)
- The Australian HIV Observational Database (AHOD)
- CHU Saint-Pierre
- University Hospital Cologne
- The EuroSIDA cohort
- Frankfurt HIV Cohort Study
- Georgian National AIDS Health Information System (AIDS HIS)
- Modena HIV Cohort
- San Raffaele Scientific Institute
- Swiss HIV Cohort Study (SHCS)
- Royal Free HIV Cohort Study
- The ATHENA national observational HIV cohort: ATHENA: AIDS Therapy Evaluation in the Netherlands
- Nice HIV Cohort
- Italian Cohort Naive Antiretrovirals (ICONA)
- PISCIS Cohort Study
- Swedish InfCare HIV Cohort
- Bonn University Hospital

SUMMARY:
The RESPOND Outcomes study is a research study around use of antiretroviral and other relevant drugs and long-term clinical outcomes in patients living with HIV. Data collected in this study will be used to answer key unanswered questions regarding treatment of people living with HIV.

DETAILED DESCRIPTION:
The specific objectives, falling into three main categories, are as follows:

1. Monitor the uptake of newer antiretroviral treatment (ART) drugs and drugs for treatment of co-infections and co-morbidities;
2. To evaluate the safety profiles of the newer individual ART drugs when used in routine clinical practice as part of either first-line or subsequent treatment regimens.
3. Investigate long term outcomes and clinical disease progression overall and in specific sub-groups

The Outcomes study is a collaboration between investigators from clinics and cohorts across Europe, Australia and South America with a willingness to share data and to use a common follow-up schedule and assessment. Participating sites have a commitment to continue to follow this large cohort that is heterogeneous in both its demographic profile and in ART prescribing patterns thus resulting in enough power to answer many key clinical questions.

The Outcomes study is a study in the RESPOND International Cohort Consortium of Infectious Diseases. RESPOND is an innovative, flexible and dynamic cohort consortium for the study of infectious diseases, including HIV, built as a generic structure for facilitating multi stakeholder involvement. In RESPOND all collected data is part of a common data repository or 'data lake', which is stored in a database located at CHIP, Rigshospitalet, Copenhagen, Denmark. Data collection in RESPOND is modular with a core data collection module onto which additional modules/studies can be added. Pseudonymised patient data can be entered manually via an online secure platform or be electronically transferred from existing local, regional or national data structures to the data lake.

In the Outcomes study data will be collected at enrolment and at annual follow-up (FU) visits. For patients living with HIV-1 enrolled and under FU, demographic, laboratory, therapeutic and clinical data on HIV and viral hepatitis will be collected once a year. Clinical event data (except AIDS other than AIDS defining malignancies) will be collected in real-time on RESPOND event forms.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed consent for the Outcomes study, if required by local/national legislation
2. Signed informed consent for the RESPOND consortium and data repository, if required by local/national legislation
3. Age ≥ 18 years of age
4. Confirmed HIV-1 infection
5. Persons receiving integrase inhibitor (INSTI) based antiretroviral therapy if have started after the later of 1/1/2012 and local cohort enrolment (i.e., during prospective follow-up in the cohort and after 1/1/2012) and have a CD4 and HIV viral load in the 12 months prior to starting INSTI or within 3 months after starting INSTI.
6. ART experienced and ART naïve persons not receiving INSTI if have a CD4 and HIV viral load in the 12 months prior to baseline or within 3 months after baseline (here, the latest of 1/1/2012 or cohort enrolment).
7. Persons lost to follow-up or who died before RESPOND enrolment should therefore still be included in the Outcomes study, provided they satisfy the other inclusion criteria.

Exclusion Criteria:

1. Persons receiving INSTI before 1/1/2012 are excluded from the Outcome study
2. Persons aged < 18 at baseline are excluded from the Outcome study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participating clinics will enrol eligible persons living with HIV. Some clinics will enrol all their eligible persons living with HIV, and others will enrol a random sample.
Sampling Method: Non-Probability Sample
Enrollment: 37853 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of HIV positive persons who initiate treatment with newer antiretroviral drugs | From date of enrolment until the date of progression, lost to follow-up or death, whichever comes first, assessed up to 6 years
  Proportion of HIV positive persons who initiate treatment with newer antiretroviral drugs and to describe changes over time in use of specific antiretroviral drugs in individual countries and diverse demographic groups
Proportion of HIV positive persons who initiate treatment of co-infections | From date of enrolment until the date of progression, lost to follow-up or death, whichever comes first, assessed up to 6 years
  Proportion of HIV positive persons who initiate treatment of co-infections and to describe changes over time in individual countries and diverse demographic groups
Proportion of HIV positive persons who initiate treatment of co-morbidities | From date of enrolment until the date of progression, lost to follow-up or death, whichever comes first, assessed up to 6 years
  Proportion of HIV positive persons who initiate treatment of co-morbidities and to describe changes over time in individual countries and diverse demographic groups
Monitor changes in plasma CD4+ T-lymphocyte counts among persons exposed to newer individual ARVs | From date of enrolment until the date of progression, lost to follow-up or death, whichever comes first, assessed up to 6 years
  Monitor changes in plasma CD4+ T-lymphocyte counts among persons exposed to newer individual ARVs
Monitor plasma HIV-RNA responses among persons exposed to newer individual ARVs | From date of enrolment until the date of progression, lost to follow-up or death, whichever comes first, assessed up to 6 years
  Monitor plasma HIV-RNA responses among persons exposed to newer individual ARVs
Evaluate the short- and long-term adverse effects of the newer ARVs when used in routine clinical practice | From date of enrolment until the date of progression, lost to follow-up or death, whichever comes first, assessed up to 6 years
  Evaluate the short- and long-term adverse effects of the newer ARVs when used in routine clinical practice as part of either first-line or subsequent treatment regimens, and whether adverse effects are reversible on discontinuation of the offending ARVs
Investigate if adverse effects are increased in some patient sub-groups in order to build clinical risk prediction scores to aid effective strategies for risk reduction | From date of enrolment until the date of progression, lost to follow-up or death, whichever comes first, assessed up to 6 years
  Investigate if adverse effects are increased in some patient sub-groups (e.g. those defined by age, gender, ethnicity, HIV-risk group, viral hepatitis- TB and other co-infections, ongoing viremia and across CD4 count strata) in order to build clinical risk prediction scores to aid effective strategies for risk reduction
Investigate if adverse effects are increased in some patient sub-groups in order to assess the risk and benefit for the individual | From date of enrolment until the date of progression, lost to follow-up or death, whichever comes first, assessed up to 6 years
  Investigate if adverse effects are increased in some patient sub-groups (e.g. those defined by age, gender, ethnicity, HIV-risk group, viral hepatitis- TB and other co-infections, ongoing viremia and across CD4 count strata) in order to assess the risk and benefit for the individual of any antiretroviral or group of antiretrovirals
Investigate long term clinical outcomes and clinical disease progression overall and in specific sub-groups | From date of enrolment until the date of progression, lost to follow-up or death, whichever comes first, assessed up to 6 years
  Investigate long term clinical outcomes and clinical disease progression overall and in specific sub-groups (e.g. those defined by age, gender, ethnicity, HIV-risk group, viral hepatitis- TB and other co-infections, ongoing viremia and across CD4 count strata)
Develop predictive risk-scores for the development of clinical outcomes to enable personalized decisions regarding risk and benefit of specific treatments in different demographic groups | From date of enrolment until the date of progression, lost to follow-up or death, whichever comes first, assessed up to 6 years
  After investigating long term clinical outcomes and clinical disease progression overall and in specific sub-groups (e.g. those defined by age, gender, ethnicity, HIV-risk group, viral hepatitis- TB and other co-infections, ongoing viremia and across CD4 count strata): to develop predictive risk-scores for the development and outcomes to enable personalized decisions regarding risk and benefit of specific treatments in different demographic groups

CONTACTS AND LOCATIONS:
Locations (18):
- The Australian HIV Observational Database (AHOD), Sydney, New South Wales, Australia
- Austrian HIV Cohort Study (AHIVCOS), Medizinische Universität Innsbruch, Innsbruck, Austria
- CHU Saint-Pierre Hospital, Brussels, Belgium
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - The EuroSIDA Study, CHIP, Rigshospitalet, Copenhagen
- Nice HIV Cohort, Centre Hospitalier Universitaire de Nice, Nice, France
- Georgian National AIDS Health Information System (AIDS HIS), IDACIRC, Tbilisi, Georgia
- Germany (3):
  - University Hospital Bonn, Bonn
  - University Hospital Cologne, Cologne
  - Frankfurt HIV Cohort Study, Goethe-University Frankfurt, Frankfurt
- Italy (3):
  - San Raffaele Scientific Institute, Ospedale San Raffaele, Milan
  - Italian Cohort Naive Antiretrovirals (ICONA), Milan
  - Modena HIV Cohort, Università degli Studi di Modena, Modena
- The ATHENA (AIDS Therapy Evaluation in the Netherlands) national observational HIV cohort, Stichting HIV Monitorin, AMC, University of Amsterdam, Amsterdam, Netherlands
- PISCIS Cohort Study, Germans Trias i Pujol University Hospital, Badalona, Spain
- Swedish InfCare HIV Cohort, Karolinska University Hospital, Stockholm, Sweden
- Swiss HIV Cohort Study (SHCS), University Hospital Zurich, Zurich, Switzerland
- Royal Free HIV Cohort Study, Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Result] Obel N, Omland LH, Kronborg G, Larsen CS, Pedersen C, Pedersen G, Sorensen HT, Gerstoft J. Impact of non-HIV and HIV risk factors on survival in HIV-infected patients on HAART: a population-based nationwide cohort study. PLoS One. 2011;6(7):e22698. doi: 10.1371/journal.pone.0022698. Epub 2011 Jul 25. PMID 21799935
- [Result] Smith CJ, Ryom L, Weber R, Morlat P, Pradier C, Reiss P, Kowalska JD, de Wit S, Law M, el Sadr W, Kirk O, Friis-Moller N, Monforte Ad, Phillips AN, Sabin CA, Lundgren JD; D:A:D Study Group. Trends in underlying causes of death in people with HIV from 1999 to 2011 (D:A:D): a multicohort collaboration. Lancet. 2014 Jul 19;384(9939):241-8. doi: 10.1016/S0140-6736(14)60604-8. PMID 25042234
- [Result] Schouten J, Wit FW, Stolte IG, Kootstra NA, van der Valk M, Geerlings SE, Prins M, Reiss P; AGEhIV Cohort Study Group. Cross-sectional comparison of the prevalence of age-associated comorbidities and their risk factors between HIV-infected and uninfected individuals: the AGEhIV cohort study. Clin Infect Dis. 2014 Dec 15;59(12):1787-97. doi: 10.1093/cid/ciu701. Epub 2014 Sep 2. PMID 25182245
- [Result] Chary A, Nguyen NN, Maiton K, Holodniy M. A review of drug-drug interactions in older HIV-infected patients. Expert Rev Clin Pharmacol. 2017 Dec;10(12):1329-1352. doi: 10.1080/17512433.2017.1377610. Epub 2017 Sep 19. PMID 28922979
- [Result] Weber R, Sabin CA, Friis-Moller N, Reiss P, El-Sadr WM, Kirk O, Dabis F, Law MG, Pradier C, De Wit S, Akerlund B, Calvo G, Monforte Ad, Rickenbach M, Ledergerber B, Phillips AN, Lundgren JD. Liver-related deaths in persons infected with the human immunodeficiency virus: the D:A:D study. Arch Intern Med. 2006 Aug 14-28;166(15):1632-41. doi: 10.1001/archinte.166.15.1632. PMID 16908797
- [Result] Kattakuzhy S, Gross C, Emmanuel B, Teferi G, Jenkins V, Silk R, Akoth E, Thomas A, Ahmed C, Espinosa M, Price A, Rosenthal E, Tang L, Wilson E, Bentzen S, Masur H, Kottilil S; ASCEND Providers. Expansion of Treatment for Hepatitis C Virus Infection by Task Shifting to Community-Based Nonspecialist Providers: A Nonrandomized Clinical Trial. Ann Intern Med. 2017 Sep 5;167(5):311-318. doi: 10.7326/M17-0118. Epub 2017 Aug 8. PMID 28785771
- [Result] Falade-Nwulia O, Suarez-Cuervo C, Nelson DR, Fried MW, Segal JB, Sulkowski MS. Oral Direct-Acting Agent Therapy for Hepatitis C Virus Infection: A Systematic Review. Ann Intern Med. 2017 May 2;166(9):637-648. doi: 10.7326/M16-2575. Epub 2017 Mar 21. PMID 28319996
- [Result] van der Meer AJ, Veldt BJ, Feld JJ, Wedemeyer H, Dufour JF, Lammert F, Duarte-Rojo A, Heathcote EJ, Manns MP, Kuske L, Zeuzem S, Hofmann WP, de Knegt RJ, Hansen BE, Janssen HL. Association between sustained virological response and all-cause mortality among patients with chronic hepatitis C and advanced hepatic fibrosis. JAMA. 2012 Dec 26;308(24):2584-93. doi: 10.1001/jama.2012.144878. PMID 23268517
- [Result] Friis-Moller N, Ryom L, Smith C, Weber R, Reiss P, Dabis F, De Wit S, Monforte AD, Kirk O, Fontas E, Sabin C, Phillips A, Lundgren J, Law M; D:A:D study group. An updated prediction model of the global risk of cardiovascular disease in HIV-positive persons: The Data-collection on Adverse Effects of Anti-HIV Drugs (D:A:D) study. Eur J Prev Cardiol. 2016 Jan;23(2):214-23. doi: 10.1177/2047487315579291. Epub 2015 Apr 16. PMID 25882821
- [Result] Mocroft A, Lundgren JD, Ross M, Fux CA, Reiss P, Moranne O, Morlat P, Monforte Ad, Kirk O, Ryom L; Data Collection on Adverse events of Anti-HIV Drugs (D:A:D) Study. Cumulative and current exposure to potentially nephrotoxic antiretrovirals and development of chronic kidney disease in HIV-positive individuals with a normal baseline estimated glomerular filtration rate: a prospective international cohort study. Lancet HIV. 2016 Jan;3(1):e23-32. doi: 10.1016/S2352-3018(15)00211-8. Epub 2015 Nov 17. PMID 26762990
- [Result] Bruyand M, Ryom L, Shepherd L, Fatkenheuer G, Grulich A, Reiss P, de Wit S, D Arminio Monforte A, Furrer H, Pradier C, Lundgren J, Sabin C; D:A:D study group. Cancer risk and use of protease inhibitor or nonnucleoside reverse transcriptase inhibitor-based combination antiretroviral therapy: the D: A: D study. J Acquir Immune Defic Syndr. 2015 Apr 15;68(5):568-77. doi: 10.1097/QAI.0000000000000523. PMID 25763785
- [Derived] Neesgaard B, Greenberg L, Miro JM, Grabmeier-Pfistershammer K, Wandeler G, Smith C, De Wit S, Wit F, Pelchen-Matthews A, Mussini C, Castagna A, Pradier C, d'Arminio Monforte A, Vehreschild JJ, Sonnerborg A, Anne AV, Carr A, Bansi-Matharu L, Lundgren JD, Garges H, Rogatto F, Zangerle R, Gunthard HF, Rasmussen LD, Necsoi C, van der Valk M, Menozzi M, Muccini C, Peters L, Mocroft A, Ryom L. Associations between integrase strand-transfer inhibitors and cardiovascular disease in people living with HIV: a multicentre prospective study from the RESPOND cohort consortium. Lancet HIV. 2022 Jul;9(7):e474-e485. doi: 10.1016/S2352-3018(22)00094-7. Epub 2022 Jun 7. PMID 35688166
- See also: The RESPOND Study — https://chip.dk/Studies/RESPOND